CLINICAL TRIAL: NCT04137744
Title: Evaluation of Axillary Reverse Mapping (ARM) in Clinically Axillary Node Negative Breast Cancer Patients
Brief Title: Axillary Reverse Mapping Using Methylene Blue Subcutaneous Injection Can Identify Arm Lymph Nodes and Vessels, Measuring Arm Size for Lymphedema, Histopathological Examination of Arm Lymph Nodes Included With Axillary Lymph Node Dissection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Hazem Nour Abdellatif, Assistant professor, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: hazem nour
Record Dates: First submitted 2019-10-21; First posted 2019-10-24 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Arm Lymphedema; Lymphatic Spread of Breast Cancer; Early Breast Cancer
Keywords: axillary reverse mapping; arm lymphedema; early breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: 2 groups of patients each 37 patient with early breast cancer one underwent ARM +ve LN biopsy with ALND, the other underwent ARM+ve LN preservation with completion of ALND
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM preservation ALND (Active Comparator): ARM +ve LN PRESERVED , ALND COMPLETED LATER ON
  Interventions: Procedure: AXILLARY REVERSE MAPPING
- conventional ALND (Active Comparator): ARM +VE NODES MARKED AND TAKEN WITH ALND
  Interventions: Procedure: AXILLARY REVERSE MAPPING

INTERVENTIONS:
Procedure: AXILLARY REVERSE MAPPING — subcutaneous injection of 1to 2 ml methylene blue 15 minutes before the procedure, identification of blue LN and lymphatic vessels
  Other Names: ALND; axillary lymph node dissection

SUMMARY:
study patients; axillary node negative breast cancer female, 74 patients randomly allocated in two groups each 37 patients , group I , where axillary reverse mapping(ARM) +ve nodes were preserved and axillary lymph node dissection completed.and group II where axillary reverse mapping +ve nodes were taken with axillary lymph node dissection(ALND) primary outcome is histopathological examination of a ARM +ve lymph nodes and volume measurements of the ipsilateral arm for development of lymphedema at 6 ,12 , and 24 months

DETAILED DESCRIPTION:
This study is comparative clinical trial carried out in the period between February 2015 and August 2019 on 74 female patients with early breast cancer. All patients were informed and signed a written consent. The study was approved from institutional review board (IRB) and ethical committee of our university.

Patient selection Patients included in the study are female patients above 18 years old, known breast cancer with clinically negative nodal metastasis who were admitted for completion ALND, after positive sentinel lymph node biopsy (SLNB).

Patients excluded from the study are those who had received chemotherapy for breast cancer, recurrent cases after conservative breast surgery, bilateral disease and pregnant cases.

Patients were randomly divided into two equal groups each 37 patients, group A; (ARM preserving ALND), where arm lymphatics and lymph nodes were identified and preserved, subsequently ALND was completed, group B; where arm lymphatics and lymph nodes were identified, marked and removed with ALND.

Technical procedures:

Axillary reverse mapping (ARM) procedure; one to two ml of methylene blue dye was subcutaneously injected in the upper medial arm in the groove between biceps muscle and triceps muscle then subsequently the area of injection was massaged for 5 minutes. During axillary dissection the (ARM) positive lymphatics and lymph nodes were identified and carefully dissected as the lymphatic vessels are very delicate, in group A the (ARM) positive lymphatics and lymph nodes were preserved and axillary clearance was completed, in group B (ARM) positive lymphatics and lymph nodes were identified, dissected, marked and taken out with ALND. The procedures were carried out with oncological surgeons familial with ALND. The limits of axillary dissection was axillary vein from above, lateral border subscapularis muscle laterally and medial border of pectoralis minor medially, long thoracic and lateral thoracic nerves were preserved intercostobrachial nerve wasn't preserved in all cases.

Data collection

* Preoperative data including demographic criteria, histopathological findings of breast biopsy and SLNB, preoperative measurement of arm volume by water displacement, circumferential measurement of the arm at the metacarpopharyngeal level, wrist level, 10 cm and 15 cm distal and proximal to the lateral epicondyle respectively.
* State of ARM positive or negative
* Follow up was carried out on outpatient clinic basis, monthly in the first 6 months then every 3 months for 2 years for data collection and later dates for regular follow up. Data was recorded including ARM histopathology (considered as the primary outcome), development of lymphedema defined as increase in arm volume by 10 % of the original size, tingling, numbness, paraesthesia and restricted shoulder movement were considered secondary outcome. Shoulder movement restriction was calculated by decrease of abduction by 10 degrees in comparison to the contralateral arm, development of local axillary recurrences, arm volume was measured at 6,12 and 24 months by water displacement method.

The collected data was properly analyzed using the proper statistical methods in SPSS 21 package.

ELIGIBILITY:
Inclusion Criteria:

* clinically free breast cancer
* sentinle LN positive

Exclusion Criteria:

* patients on chemotherapy for breast cancer
* recurrent cases after conservative breast surgery
* bilateral disease and pregnant cases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female , early breast cancer
Enrollment: 74 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
histopathologic examination of ARM +ve LN | IMMEDIATE POSTOPERATIVE
  EITHER +VE OR -VE
ARM LYMPHOEDEMA | 2 years postoperative
  INCREASE OF THE ARM VOLUME BY 10%

SECONDARY OUTCOMES:
restriction of shoulder movement | 2 years
  in comparison to the other side

CONTACTS AND LOCATIONS:
Overall Officials: hazem nour, MD, Principal Investigator — assistant professor, general surgery
Locations (1):
- Zagazig Faculty of Medicine, Zagazig, Sharqya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided